CLINICAL TRIAL: NCT05721521
Title: The Effects of Exercise Intensity on Mood and Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Katie Barfoot, Principal Investigator, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2022-133-KB
Record Dates: First submitted 2022-12-12; First posted 2023-02-10 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Healthy; Exercise; Mood
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High intensity (Experimental)
  Interventions: Other: Spin Bike Exercise
- Moderate intensity (Experimental)
  Interventions: Other: Spin Bike Exercise
- Low intensity (Experimental)
  Interventions: Other: Spin Bike Exercise
- No exercise (control) (Placebo Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Spin Bike Exercise — 30 minute spin bike class led by a qualified instructor.
  Arms: High intensity; Low intensity; Moderate intensity
Other: Control — 30 minute completing seated activities (e.g., wordsearches)
  Arms: No exercise (control)

SUMMARY:
The study will adopt a between-within group design where participants will exercise at 1 of 4 intensities for 30 minutes at SportsPark Reading. Mood, mental health (e.g., state anxiety and immediate depressive feelings) and physiological parameters (heart rate, blood pressure and body temperature) will be assessed before and after exercise intervention to compare the acute change across time for each intensity condition (no exercise (control), low, moderate, high).

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years old

Exclusion Criteria:

* If participants' General Practitioner (GP) has advised them against exercising at low, moderate or high intensities
* Recent injuries within the last 12 weeks
* Physical health conditions that may be affected by exercising (e.g., asthma)
* Taking blood pressure medications

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline state anxiety | In the immediate 10 minutes after the end of the intervention
  State subscale of the State-Trait Anxiety Inventory (STAI-S). The State-Trait Anxiety Inventory (STAI) measures both state and trait anxiety in adults; it can be used to distinguish whether individuals are experiencing anxiety. Trait anxiety refers to the participant's disposition to anxiety, whereas state anxiety measures the current anxiousness of participants and is more labile. STAI is a questionnaire consisting of forty self-report items. Subjects are asked to rate the intensities of anxious feelings on a four-point scale: not at all, somewhat, moderately so or very much so. Scores range from twenty to eighty, where higher scores correlate with higher state or trait anxiety.
Change from baseline current mood | In the immediate 10 minutes after the end of the intervention
  Positive and Negative Mood Schedule (PANAS). This questionnaire contains 20 items consisting of 10 positive and 10 negative emotions. The participants indicate to what extent they feel each emotion right now on a 5-point Likert Scale of 'very slightly =1 or not at all' to 'Extremely= 5'. Adding up the total positive and negative scores will produce overall positive and negative mood scores.

SECONDARY OUTCOMES:
Change from baseline depressive aspects of mood | In the immediate 10 minutes after the end of the intervention
  Immediate Mood Scaler (IMS). This questionnaire contains 22 items developed to assess dynamic components of mood. Participants are asked to rate their current mood state on a continuum using 7-point Likert scales (e.g., happy-sad, distracted-focused, sleepy-alert). For each item, an integer score between 1 and 7 is derived. The total score for this scale is the sum of the scores on all 22 items, where a higher score is indicative of better mood.

OTHER OUTCOMES:
Change from baseline blood pressure | In the immediate 10 minutes after the end of the intervention
Change from baseline temperature | In the immediate 10 minutes after the end of the intervention
Change from baseline heart rate | approx. 1 hour in total
  Measured by a chest strap heart rate monitor
Change from baseline stress appraisal of intervention | In the immediate 10 minutes after the end of the intervention
  The stress appraisal questionnaire captures 1) perceived situational and personal demands, and 2) personal resources. To the extent that perceived demands outweigh resources then individuals are anticipated to be in a "threat" state, whereas when resources outweigh demands individuals are expected to be in a "challenge" state.
  A questionnaire is given pre-task that captures stress appraisals after knowledge of the task is obtained but before the task itself. There is a post-task questionnaire that assesses individuals' perceptions of the demands and resources after the task.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom